CLINICAL TRIAL: NCT00999583
Title: High Dose of Erythropoietin Analogue After Cardiac Arrest: a Multicentre, Randomised, Controlled Trial (Epo-ACR-02 Trial)
Brief Title: High Dose of Erythropoietin Analogue After Cardiac Arrest
Acronym: Epo-ACR-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P071217
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Comatose Survivors of Cardiac Arrest
Keywords: Cardiac arrest; erythropoietin; post-anoxic encephalopathy; neuroprotective drugs
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPO (Experimental): five injections maximum of 40000 UI EPO
  Interventions: Drug: EPOETINE ALPHA
- Control (Active Comparator): Classical take care
  Interventions: Other: Control arm

INTERVENTIONS:
Drug: EPOETINE ALPHA — 5 injections of 40000 UI of EPO
  Arms: EPO
Other: Control arm — Usual take care of cardiac arrest
  Arms: Control

SUMMARY:
The investigators hypothesised that the neuroprotective effects of erythropoietin and its analogues could lead to an improve outcome after cardiac arrest. To test this hypotheses, the investigators designed a randomized, multicentre, simple blind trial in which all participating patients will be receive usual treatments and 50% of them will also receive a high dose of epoetin alpha (an analogue of erythropoietin) in an "add on" fashion. The main end point will be the proportion of patients in each arm who will reach at day 60 the best level of recovery, using a 5 level score.

DETAILED DESCRIPTION:
Rationale:

A recent pilot study showed encouraging results regarding the potentially beneficial effects of high dose epoetin alpha (an analogue of erythropoietin) when administered early after cardiac arrest. In this open label and non randomized trial, a high proportion of patients survived without significant cerebral disability and without experiencing severe adverse events (CARIOU et al. Resuscitation 2008). Efficiency of this treatment should now be evaluated in a randomized trial.

Hypotheses:

An early administration of a high dose of epoetin alpha (Epo) after cardiac arrest resuscitation could improve the neurological outcome of these patients by comparison with standard treatment. The proportion of patients reaching the level 1 of the Pittsburgh CPC scale (i.e., no or minor cerebral disability) at day 60 could attain 45% in the interventional group versus 30% as expected in the control group.

Design:

Multicentre, randomised, controlled, simple blind trial ("add on study").

Main goal:

To test the efficiency of a high dose of Epo administered at the early stage of the post-cardiac arrest period regarding its ability to improve the neurological outcome of these patients, when compared with standard care (including hypothermia when indicated).

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 80
* Witnessed out-of-hospital cardiac arrest, presumed of cardiac origin (non asphyxic)
* Time from cardiac arrest and recovery of circulatory activity less than 60 minutes
* Persistent coma after ROSC (Coma Glasgow Scale < 7)

Exclusion criteria:

* Out-of-hospital cardiac arrest with evidence of extra-cardiac cause (trauma, sepsis, acute respiratory insufficiency, asphyxia)
* Previous or chronic treatment with erythropoietin or analogues
* Pregnancy
* Rapidly fatal underlying disease (expected life duration < 6 months)
* No social security

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2009-10; Primary Completion 2013-07 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of patients reaching a CPC (cerebral performance category) level 1 in each group | at day 60

SECONDARY OUTCOMES:
Distribution of patients in CPC (cerebral performance category) scale | at day 30 and day 60
ICU, hospital D30 and D60 mortality | during hospitalization and at day 30 and day 60
All adverse events (including thrombotic events) | until day 60

CONTACTS AND LOCATIONS:
Overall Officials: Alain Cariou, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Medical intensive care unit of Cochin-St Vincent de Paul university Hospital, Paris, France

REFERENCES:
- [Result] Cariou A, Deye N, Vivien B, Richard O, Pichon N, Bourg A, Huet L, Buleon C, Frey J, Asfar P, Legriel S, Narcisse S, Mathonnet A, Cravoisy A, Dequin PF, Wiel E, Razazi K, Daubin C, Kimmoun A, Lamhaut L, Marx JS, de la Garanderie DP, Ecollan P, Combes A, Spaulding C, Barat F, Ben Boutieb M, Coste J, Chiche JD, Pene F, Mira JP, Treluyer JM, Hermine O, Carli P; Epo-ACR-02 Study Group. Early High-Dose Erythropoietin Therapy After Out-of-Hospital Cardiac Arrest: A Multicenter, Randomized Controlled Trial. J Am Coll Cardiol. 2016 Jul 5;68(1):40-9. doi: 10.1016/j.jacc.2016.04.040. PMID 27364049
- [Derived] Nishiwaki H, Abe Y, Suzuki T, Hasegawa T, Levack WM, Noma H, Ota E. Erythropoiesis-stimulating agents for preventing acute kidney injury. Cochrane Database Syst Rev. 2024 Sep 20;9(9):CD014820. doi: 10.1002/14651858.CD014820.pub2. PMID 39301879
- [Derived] Madelaine T, Cour M, Roy P, Vivien B, Charpentier J, Dumas F, Deye N, Bonnefoy E, Gueugniaud PY, Coste J, Cariou A, Argaud L. Prediction of Brain Death After Out-of-Hospital Cardiac Arrest: Development and Validation of the Brain Death After Cardiac Arrest Score. Chest. 2021 Jul;160(1):139-147. doi: 10.1016/j.chest.2021.01.056. Epub 2021 Jun 8. PMID 34116828
- [Derived] Boissady E, Kohlhauer M, Lidouren F, Hocini H, Lefebvre C, Chateau-Jouber S, Mongardon N, Deye N, Cariou A, Micheau P, Ghaleh B, Tissier R. Ultrafast Hypothermia Selectively Mitigates the Early Humoral Response After Cardiac Arrest. J Am Heart Assoc. 2020 Dec;9(23):e017413. doi: 10.1161/JAHA.120.017413. Epub 2020 Nov 17. PMID 33198571